CLINICAL TRIAL: NCT00402220
Title: A Double-blind Sham Controlled Trial of rTMS in Treatment Resistant Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fitzgeraldp
Record Dates: First submitted 2006-11-18; First posted 2006-11-22 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): active TMS
  Interventions: Drug: TMS
- 2 (Placebo Comparator): Sham TMS
  Interventions: Device: Sham TMS

INTERVENTIONS:
Drug: TMS — Active Transcranial Magnetic Stimulation
  Arms: 1
Device: Sham TMS — Sham Transcranial Magnetic Stimulation
  Arms: 2

SUMMARY:
The main treatment option for Treatment Resistant Depression is electroconvulsive therapy (ECT) which is often effective but complicated by cognitive side effects, need for anaesthesia and considerable stigma.

In recent years considerable efforts have been made to increase public awareness about depression and increase access to services. However, the increasing number of patients accessing treatment for depression in clinical services is also likely to be accompanied by a sizeable increase in the number of patients with TRD. Despite the demand, relatively few treatment options are available to such patients. One of the only substantially new treatments developed for TRD in recent years has been the advent of repetitive transcranial magnetic stimulation (rTMS). Repetitive TMS has been evaluated in over 20 trials conducted over the last 10 years. Previous research indicates that rTMS has antidepressant activity; however, the proportion of patients who respond to rTMS and the degree of treatment response demonstrated in trials to date is limited. The limitations of these studies include relatively small samples and limited duration of treatment (i.e., 2 weeks) as well as a lack of long term follow-up. As rTMS is gradually entering use in routine clinical practice (for example, recent regulation of its use in Canada), research is urgently required to establish ways to enhance treatment response both in regards to the extent of response within individuals and the proportion of individuals in whom rTMS has effects.

Stimulation site is another important treatment factor; thus far almost all of the trials of rTMS in TRD conducted have evaluated the utility of high frequency left prefrontal cortex (PFC) rTMS (HFL-TMS). In addition, several studies have evaluated the treatment efficacy of low frequency rTMS to right PFC (LFR-TMS). In a previously published study we have demonstrated that these two approaches have similar therapeutic benefit and both were superior to sham stimulation.

A promising new approach to enhance efficacy involves combining LFR-TMS and HFL-TMS in a sequential manner. We describe this as sequential bilateral rTMS (SB-rTMS). We have recently published the results of the first substantial evaluation of SB-rTMS showing not only a superiority to placebo in TRD but also a therapeutic response that is substantially superior to response rates in most of the published studies of unilateral rTMS (>50% of patients achieving standard criteria for clinical response compared to usually <30% in most studies). In this proposed research study, we will directly test the hypothesis that SB-rTMS produces a greater therapeutic response than HFL-TMS and compare both of these forms of stimulation to placebo (i.e., sham) stimulation.

DETAILED DESCRIPTION:
Justification for project

TRD is clearly a major health issue - depression is common, results in marked morbidity and mortality and a large percentage of patients do not respond to, or cannot tolerate standard treatment. The development of new treatments for this condition is undoubtedly required. International efforts are underway to try and establish the efficacy of HFL-TMS to the point where the technique may be approved by regulatory authorities and clinically introduced. However, clearly the response rate to HFL-TMS is suboptimal for its widespread use.

The overall goal of this research program is to develop rTMS methods to the point at which they are highly relevant and applicable to clinical practice. None of the substantial international studies is focusing on novel applications such as SBrTMS. As an outcome, we expect positive results to change the focus of rTMS application and practice nationally and internationally. If we can follow our well received initial study of this technique with a substantial comparative trail as planned here, it will provide enough evidence for the more widespread adoption and testing of SBrTMS as a viable alternative to HFL-TMS. Ultimately, this or a modification of it, may become the rTMS administration method of choice.

Additionally, we will have a sufficient sample size to start to explore meaningful predictors of clinical response including biological, psychosocial/personality variable predictors.

Hypotheses / Research Questions

Primary Hypothesis

* Hypothesis 1: Treatment with left sided and SBrTMS will both result in a greater reduction in HAMD and MADRS scores than sham rTMS.
* Hypothesis 2: Treatment with SBrTMS will result in a greater reduction in HAMD and MADRS scores than left sided rTMS applied alone.

Secondary Hypotheses

• Greater than 50% of treatment responders to rTMS will continue to experience clinical benefits from rTMS, as indexed by persistently low HAMD and MADRS scores, at 6 months post acute treatment.

Methodology including project design and sequence of procedures

Experimental Design

The study will involve a 2 phases of treatment: an acute treatment phase of 3-9 weeks duration and a maintenance treatment phase, lasting 52 weeks. In the initial 3 weeks of the acute treatment phase the study will be randomised, double blind and sham-controlled with three arms:

1. SBrTMS
2. Unilateral left rTMS
3. Sham rTMS

Prior to randomization, participants will undergo an EEG and MRI (see below for more detail). The EEG and MRI will be repeated once during the active treatment phase.

Randomization will occur via the generation of a single computer number sequence. Subjects will be randomised immediately prior to the commencement of the first treatment session, after the measurement of bilateral resting motor thresholds with standard means [30].

Acute treatment will be administered daily, 5 days per week initially for three weeks (i.e. 15 treatments). Following 3 weeks of treatment response will be assessed and the blind broken. At this point non responders (i.e. HAM-D score > 10) who have been receiving active treatment will be offered an additional 3 weeks of treatment at the same treatment parameters. Responders who have been receiving active treatment will enter the maintenance phase. At week 6 treatment response will again be assessed and non responders will be offered a final 3 weeks of active treatment while responders will enter the maintenance phase. At week 9 response will again be assessed and non responders will cease their participation in the trial, while responders will continue onto the maintenance phase. With regard to the sham treatment arm, subjects who respond to treatment and received sham treatment will be discontinued from the study at week 3. Those subjects who are classified as non responders and were in the sham treatment arm will be randomised to one of the two active treatment arms and receive an additional 3 weeks of active treatment.

The maintenance phase will be open labeled and consist of weekly treatments at the same parameters to which patients initially responded, for a total of 8 weeks. Maintenance treatment will then be further reduced to fortnightly treatments for 44 weeks. Patients will be evaluated clinically every 2 weeks. Should patients relapse (i.e. a HAM-D score of >15 for 2 consecutive weeks), they will be offered active treatment only (i.e. no sham treatment) for up to six weeks at the same stimulus parameters to which they previously experienced a response.

Subjects

Inclusion Criteria: Patients will be included if they:

1. Have a DSM-IV diagnosis of a major depressive episode (SCID 11).
2. Aged 18-85.
3. Have treatment resistant depression at Stage II of the Thase and Rush classification [31]; .e. have failed to achieve a clinical response, or did not tolerate, at least two separate antidepressant trials of sufficient dose for at least 6 weeks.
4. Have a Hamilton Depression Rating Scale Score of > 20 (moderate - severe depression). Including only a severely ill group of subjects limits the placebo response rate [32]. Moreover, this will allow us to address the application of rTMS methods in the most clinically relevant subgroup of patients (in addition helping to constrain group heterogeneity, a major issue in depression research).
5. Have had no increase or initiation of new antidepressant (or other psychoactive) therapy in the 4 weeks prior to screening.

Additional Exclusion Criteria:

1. Patients who have an unstable medical condition, neurological disorder or any history of a seizure disorder or are currently pregnant or lactating.
2. In the opinion of the investigator, are a sufficient suicidal risk to require immediate electro-convulsive therapy.
3. Have a current DSM IV diagnosis of substance abuse or dependence disorder, a diagnosis of a personality disorder (SCID II) or another axis 1 disorder.

Please note: several of these criteria (e.g. inclusion criteria 1 & 2, exclusion criteria 3) have been selected to explicitly constrain the heterogeneity of the sample to increase the likely power of the study to detect differences between the groups given the potentially subtle difference between the treatment methods.

Sample Size Calculations We aim to recruit 40 patients into each group (total n=120). The sample size calculation for the study was conducted based on the within group standard deviation of 12.9 (this was the standard deviation for baseline to final study visit in our SBrTMS study) and between group difference of 5.0 points. With an alpha of 0.05 the study will have a power of 0.87 to detect a difference in end scores between the 3 groups (calculation in PASS 8.0).

Clinical Measures Demographic variables and potential co-variates will be recorded at baseline following a clinical interview. These will include the duration of the current episode, years from first diagnosis, number of previous episodes, type and dose of current and previous treatment and family history of mood disorder.

Clinical measures will be performed at randomization, at 3 and 6 weeks (and 9 weeks in the patients in the extension phase) as well as at the follow up assessments. A trained rater who is blind to treatment type will administer all measures. Raters will be required to maintain >90% reliability on the primary outcome assessments on ratings with 6 monthly assessments based on videotaped interviews.

To ensure comparability with previous studies, the primary outcome variable will be the 17-item Hamilton Rating Scale for Depression (HAMD). Other outcome measures will include the Montgomery-Asberg Depression Rating Scale (MADRS), Beck Depression Questionnaire (BDI), Brief Psychiatric Rating Scale (BPRS) and an interview to record the subjective experiences of TMS and any adverse events. Final response and remission rates will be measured using standard rating scale score criteria but the patients will need to achieve these scores at the study end and at the 2 week follow up assessment.

Assessments made at baseline to explore potential predictors of clinical response will include the CORE rating of melancholia [33], the Measure of Parental Styles [34], the Depressive Personality Inventory [35] and the Costello and Comrey trait anxiety measure [36].

A battery of cognitive tests will be administered prior to commencement and at 3, 6 and 9 weeks in the active treatment phase with a specific focus on attention and memory:

HVLT, Controlled oral word association, Trail making A&B, Digit Span The inclusion of these measures in the will assess the potential beneficial effects of TMS on frontally mediated cognitive functions as well as act as a safety check.

TMS Treatment TMS will be administered with a Medtronic Magpro30 magnetic stimulator using a 70mm figure of 8 coil. Prior to the commencement of treatment TMS, single pulse TMS will be used to measure the resting motor thresholds (RMT) for the abductor pollicis brevis (APB) bilaterally in all subjects using standard published methods [30].

Stimulation parameters rTMS will be administered on a daily basis 5 days per week for all subjects:

Bilateral:

Left: 10Hz, 100% RMT, 30 Trains, 5 second duration, 25 second inter-train interval Right: 1 Hz, 100% RMT, 1 Train of 600 pulses

Left Unilateral:

Left: 10Hz, 100% RMT, 30 Trains, 5 second duration, 25 second inter-train interval Right: as above, BUT, applied with a Medtronic sham coil Sham: the following applied with a sham coil Left: 10Hz, 100% RMT, 30 Trains, 5 second duration, 25 second inter-train interval Right: 1 Hz, 100% RMT, 1 Train of 600 pulses Missed sessions will be 'made up' by an extension of the treatment duration but only one missed session will be allowed weekly and only one missed session in a row.

Stimulation localisation This will follow standard procedures. Firstly, the site for the optimal activation of the abductor pollicis brevis muscle in the contralateral hand will be located whilst stimulating the relevant motor cortical region at supra-threshold intensity. This site will be marked on the scalp. We will then measure 6 cm anteriorly on the scalp surface and mark it with ink. This point will be then used as the site of stimulation. The majority of rTMS studies have measured 5 cm anteriorly. However, this has been shown to result consistently in localisation that is posterior to the dorsolateral PFC [37]. The measurement described here should result in more consistent treatment of dorsolateral PFC but still provide considerable stimulation overlap with the established '5 cm' site.

Imaging MRI imaging will be conducted before the commencement of treatment (all subjects) and at the end of the active treatment phase where possible. Each subject will undergo a 3D sagittally orientated T1 weighted structural MR scan on the 1.5 Tesla MRI scanner at the Alfred (128 slices). Analysis of scalp to cortex distance in prefrontal cortex and at the site of stimulation will be conducted using previously published methods. This will allow the post hoc analysis of the relationship between scalp to cortex distance and treatment response. In addition, where possible subjects will undergo additional measures of white matter tract integrity (diffusion tensor imaging) and activation. None of the scanning procedures will involve the administration of contrast.

Electroencephalography (EEG) EEG before and after the acute phase of treatment will be used to examine mean absolute spectral power within 5 frequency bands. The mean absolute power (in squared microvolts per hertz) will then be computed within the following 5 frequency bands: delta (0.5-3.5 Hz), theta (3.5-7.5 Hz); alpha (7.5-12.5 Hz); beta 1 (12.5-20.5 Hz), and beta 2 (20.5-32.5 Hz). EEG activation / spectral power will be assessed at rest (eyes open and closed) and during cognitive engagement in several tasks.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they:

1. Have a DSM-IV diagnosis of a major depressive episode (SCID 11).
2. Aged 18-85.
3. Have treatment resistant depression at Stage II of the Thase and Rush classification [31]; .e. have failed to achieve a clinical response, or did not tolerate, at least two separate antidepressant trials of sufficient dose for at least 6 weeks.
4. Have a Hamilton Depression Rating Scale Score of > 20 (moderate - severe depression). Including only a severely ill group of subjects limits the placebo response rate [32]. Moreover, this will allow us to address the application of rTMS methods in the most clinically relevant subgroup of patients (in addition helping to constrain group heterogeneity, a major issue in depression research).
5. Have had no increase or initiation of new antidepressant (or other psychoactive) therapy in the 4 weeks prior to screening.

Exclusion Criteria:

1. Patients who have an unstable medical condition, neurological disorder or any history of a seizure disorder or are currently pregnant or lactating.
2. In the opinion of the investigator, are a sufficient suicidal risk to require immediate electro-convulsive therapy.
3. Have a current DSM IV diagnosis of substance abuse or dependence disorder, a diagnosis of a personality disorder (SCID II) or another axis 1 disorder.

Please note: several of these criteria (e.g. inclusion criteria 1 & 2, exclusion criteria 3) have been selected to explicitly constrain the heterogeneity of the sample to increase the likely power of the study to detect differences between the groups given the potentially subtle difference between the treatment methods.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The 17- item Hamilton Rating Scale for Depression (HAM-D) | every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Fitzgerald, MBBS, MPM, PhD, FRANZCP, Principal Investigator — Alfred Psychiatry Research Centre
Locations (1):
- Alfred Psychiatry Research Centre, Prahran, Victoria, Australia